CLINICAL TRIAL: NCT06046040
Title: Phase I, Open-Label Study of Dually Armored Chimeric Antigen Receptor (CAR) T Cells (TmPSMA-02) in Patients With Metastatic Castrate-Resistant Prostate Cancer (mCRPC)
Brief Title: TmPSMA-02 in mCRPC
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Prostate Cancer Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 11823
Record Dates: First submitted 2023-09-13; First posted 2023-09-21 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Castrate-Resistant Prostate Cancer (mCRPC)

STUDY DESIGN:
Intervention Model Description: This is a Phase I, open-label dose finding study to assess the safety, tolerability, manufacturing feasibility, and preliminary efficacy of TmPSMA-02 CAR T cells in patients with metastatic castrate-resistant prostate cancer (mCRPC). Up to 4 total dose levels will be evaluated using a 3+3 dose escalation design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dose Level -1 (Experimental): After lymphodepleting chemotherapy subjects to receive 1x10(7) TmPSMA-02 CAR T Cells
  Interventions: Drug: TmPSMA-02 CAR T Cells
- Dose Level 1 (Experimental): After lymphodepleting chemotherapy subjects to receive 5 x10(7) TmPSMA-02 CAR T Cells
  Interventions: Drug: TmPSMA-02 CAR T Cells
- Dose Level 2 (Experimental): After lymphodepleting chemotherapy subjects to receive 1x10(8) TmPSMA-02 CAR T Cells
  Interventions: Drug: TmPSMA-02 CAR T Cells
- Dose Level 3 (Experimental): After lymphodepleting chemotherapy subjects to receive 3x10(8) TmPSMA-02 CAR T Cells
  Interventions: Drug: TmPSMA-02 CAR T Cells

INTERVENTIONS:
Drug: TmPSMA-02 CAR T Cells — TmPSMA-02 CAR T cells: autologous T cells transduced with a lentiviral vector to express an anti-PSMA CAR containing a humanized J591-derived scFv and CD2 co-stimulatory domain, and dually armored with a TGFβRDN and PD1.CD28 switch receptor.

SUMMARY:
This is a Phase I, open-label dose finding study to assess the safety, tolerability, manufacturing feasibility, and preliminary efficacy of TmPSMA-02 CAR T cells in patients with metastatic castrate-resistant prostate cancer (mCRPC). Up to 4 total dose levels will be evaluated using a 3+3 dose escalation design.

DETAILED DESCRIPTION:
This is a Phase I, open-label dose finding study to assess the safety, tolerability, manufacturing feasibility, and preliminary efficacy of TmPSMA-02 CAR T cells in patients with metastatic castrate-resistant prostate cancer (mCRPC). Up to 4 total dose levels will be evaluated using a 3+3 dose escalation design as described below. Dose escalation will begin with Dose Level 1 as follows:

* Dose Level 1 (N = 3 to 6): Subjects will receive a single dose of 5 x 107 TmPSMA-02 CAR T cells via IV infusion administration on Day 0, following lymphodepletion with fludarabine and cyclophosphamide. This dose level will be evaluated as follows:

  * If 1 DLT/3 subjects occurs, the study will enroll an additional 3 subjects at this dose level.
  * If 0 DLT/3 subjects or 1 DLT/6 subjects occur, the study will advance to Dose Level 2 (DL2).
  * In the event that 2 or more DLTs occur at Dose Level 1 (DL1), enrollment at this dose level will be stopped and Dose Level -1 (DL-1) will be opened. In Dose Level -1, subjects will receive a de-escalated dose of 1 x 107 TmPSMA-02 CAR T cells following lymphodepletion.

If 0 DLT/3 or 1 DLT/3 subjects occurs at DL-1, the study will enroll an additional 3 subjects at this dose level.

If ≥ 2 DLTs occur at any time, enrollment at this dose level will be stopped.

Dose Level 2 (N = 3 to 6): Subjects will receive a single fixed dose of 1 x 108 TmPSMA-02 CAR T cells via IV infusion on Day 0, following lymphodepletion with fludarabine and cyclophosphamide. This dose level will be evaluated as follows:

* If 1 DLT/3 subjects occurs, the study will enroll an additional 3 subjects at this dose level.
* If 0 DLT/3 subjects or 1 DLT/6 subjects occur, the study will advance to Dose Level 3 (DL3).
* If 2 DLTs occur at any time, enrollment at this dose level will be stopped. If less than 6 subjects were treated at the previous dose level (DL1), additional subjects will be enrolled at that dose level to reach a minimum of 6 DLT-evaluable subjects for MTD determination.

  • Dose Level 3 (N = 3 to 6): Subjects will receive a single fixed dose of 3 x 108 TmPSMA-02 CAR T cells via IV infusion Day 0, following lymphodepletion with fludarabine and cyclophosphamide. This dose level will be evaluated as follows:
* If 1 DLT/3 subjects occurs, the study will enroll an additional 3 subjects at this dose level.
* If 0 DLT/3 subjects occurs, the study will still enroll an additional 3 subjects at this dose level to allow for MTD determination.
* If 2 DLTs occur at any time, enrollment at this dose level will be stopped. If less than 6 subjects were treated at the previous dose level (DL2), additional subjects will be enrolled at that dose level to reach a minimum of 6 DLT-evaluable subjects for MTD determination.

The highest dose at which 0 or 1 DLT occurs in 6 DLT-evaluable subjects will be declared the MTD.

Retreatment Infusions:

The Retreatment Phase will remain closed until sufficient safety and persistence data is available in initial subjects, and DSMB and FDA approval to open Retreatment has been received.

Subjects who have demonstrated clinical benefit after their initial TmPSMA-02 CAR T cell infusion (e.g., minimum disease response of stable disease, etc.) may also be eligible to receive retreatment with TmPSMA-02 CAR T cells at the physician-investigator's discretion. The TmPSMA-02 retreatment dose administered must either be a) the CAR T cell dose that the subject previously received without DLTs, or b) a CAR T cell dose that is less than or equal to a dose level that has been evaluated for safety in ≥ 3 other subjects without evidence of DLTs. As retreatment infusions will not be used for formal DLT assessments/MTD determination, there are no protocol-defined staggering requirements.

ELIGIBILITY:
Inclusion Criteria:

1. Signed, written informed consent
2. Adult participants ≥ 18 years of age
3. Metastatic castrate-resistant prostate cancer (mCRPC)
4. Castrate levels of testosterone (<50 ng/dL) with/without the use of androgen-deprivation therapy
5. Received at least one prior standard therapy for systemic treatment in the mCRPC setting, including at least one second generation androgen receptor signaling inhibitor (e.g., enzalutamine, apalutamide, darolutamide, or abiraterone) or a taxane-based regimen (e.g., docetaxel, cabazitaxel, etc).
6. Adequate organ function within 4 weeks of eligibility confirmation by a physician-investigator defined as:

   1. Serum creatinine ≤ 1.5 mg/dl or creatinine clearance ≥ 50 cc/min per the Cockcroft-Gault Equation; Patient must not be on dialysis
   2. ALT/AST ≤ 3 x ULN
   3. Serum total bilirubin ≤ 1.5 mg/dL, unless the subject has Gilbert's syndrome (if so, serum total bilirubin must be ≤3.0 mg/dL)
   4. Left Ventricle Ejection Fraction (LVEF) ≥ 45% confirmed by ECHO
   5. Must have a minimum level of pulmonary reserve defined as ≤ Grade 1 dyspnea and pulse oxygen > 92% on room air
7. Patients must have adequate hematologic reserve within 4 weeks of eligibility confirmation by a physician-investigator and must not be dependent on transfusions to maintain these hematologic parameters. Adequate hematologic reserve is defined as:

   1. Hemoglobin ≥ 8 g/dL
   2. Absolute neutrophil count ≥ 1000/μL
   3. Platelet count ≥ 75,000/μL
8. ECOG Performance Status that is either 0 or 1.
9. Patients who have not undergone bilateral orchiectomy must be able to continue GnRH therapy during the study.
10. Participants of reproductive potential must agree to use acceptable birth control methods, as described in the protocol.

Exclusion Criteria:

1. Active hepatitis B or hepatitis C infection
2. Any other active, uncontrolled infection
3. Class III/IV cardiovascular disability according to the New York Heart Association Classification.
4. Severe, active co-morbidity that in the opinion of the physician-investigator would preclude participation in the study.
5. Active invasive cancer, other than the proposed cancer included in the study, within 2 years prior to eligibility confirmation by a physician-investigator. [Note: non-invasive cancers treated with curative intent (e.g., non-melanoma skin cancer) may still be eligible].
6. Patients requiring chronic treatment systemic steroids or immunosuppressant medications. Low-dose physiologic replacement therapy with corticosteroids equivalent to prednisone 10 mg/day or lower, topical steroids and inhaled steroids are acceptable. For additional details regarding use of steroid and immunosuppressant medications, please see Section 5.6.
7. Prior treatment with autologous T-cell therapy, with the exception of Sipuleucel-T.
8. Prior allogeneic stem cell transplant.
9. Active autoimmune disease requiring systemic immunosuppressive treatment equivalent to ≥ 10mg of prednisone. Patients with autoimmune neurologic diseases (such as MS) will be excluded.
10. History of allergy or hypersensitivity to study product excipients (human serum albumin, DMSO, and Dextran 40).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-01-31 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2042-01-31 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with dose limiting toxicities (DLTs) | 28 days after TmPSMA-02 CAR T cell infusion
Determination of maximum tolerated dose (MTD) | 28 days after TmPSMA-02 CAR T cell infusion
Incidence of Adverse Events as assessed by CTCAE v5.0 | Up to 15 years

SECONDARY OUTCOMES:
Percentage of manufacturing products that meet release criteria | Up to 3 years
Overall Response Rate (ORR) | Up to 3 months
Duration of Response (DOR) | up to one year
Progression Free Survival (PFS) | Up to one year
Overall Survival (OS) | Up to one year
Percent Change in PSA from Baseline | Up to one year

CONTACTS AND LOCATIONS:
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Wang Y, Zhao G, Wang S, Li N. DNTGF-betaR armored CAR-T cell therapy against tumors from bench to bedside. J Transl Med. 2024 Jan 11;22(1):45. doi: 10.1186/s12967-023-04829-6. No abstract available. PMID 38212769